CLINICAL TRIAL: NCT02905292
Title: Inactivity, Balance Problems and Fall Risk in Institutionalized Frail Elderly: What is the Impact of Benign Paroxysmal Positional Vertigo (BPPV) and Treatment Effectiveness?
Brief Title: Inactivity, Balance Problems and Fall Risk in Institutionalized Frail Elderly
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hasselt University (Other)
Responsible Party: Principal Investigator, JSpildooren, dr., Hasselt University
Other Study IDs: BPPV-ELDERLY-001
Record Dates: First submitted 2016-09-14; First posted 2016-09-19 (Estimated); Last update posted 2016-09-19 (Estimated); Status verified 2016-09

CONDITIONS: Institutional Frail Elderly

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: evaluation and treatment maneuver for BPPV

SUMMARY:
The overall objective of the research is to identify the prevalence and incidence of BPPV and the impact on balance problems, fall risk and inactivity in frail elderly. The investigators will demonstrate the importance of early diagnosis and treatment in this patient group.

ELIGIBILITY:
Inclusion Criteria:

* Institutionalized in a nursing home for at least 3 months
* Able to understand and follow simple instructions
* Able to stand independently for 30 seconds
* Willing to participate in the study

Exclusion Criteria:

* diagnosis of progressive neurological diseases (such as Amyotrophic Lateral Sclerosis) resulting in a fast decline within 3 months
* Rehabilitating for a neurological or orthopaedic incident such as knee prosthesis, stroke,… )
* Contra-indication for Hallpike and Epley maneuver

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: institutionalized frail elderly
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-06 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
outcome of the vestibular bedside testing | baseline
  outcome of the vestibular bedside testing (i.e. Dix-Hallpike-, side lying- or roll-test)
outcome of the vestibular bedside testing | month 1
  outcome of the vestibular bedside testing (i.e. Dix-Hallpike-, side lying- or roll-test)
outcome of the vestibular bedside testing | month 2
  outcome of the vestibular bedside testing (i.e. Dix-Hallpike-, side lying- or roll-test)
outcome of the vestibular bedside testing | month 3
  outcome of the vestibular bedside testing (i.e. Dix-Hallpike-, side lying- or roll-test)
outcome of the vestibular bedside testing | month 4
  outcome of the vestibular bedside testing (i.e. Dix-Hallpike-, side lying- or roll-test)
outcome of the vestibular bedside testing | month 5
  outcome of the vestibular bedside testing (i.e. Dix-Hallpike-, side lying- or roll-test)
outcome of the vestibular bedside testing | month 6
  outcome of the vestibular bedside testing (i.e. Dix-Hallpike-, side lying- or roll-test)
static and dynamic balance using the Mobility lab (APDM-sensors) | baseline
  static and dynamic balance using the Mobility lab (APDM-sensors): iSway (COP sway area and velocity with and without vision), iTUG
static and dynamic balance using the Mobility lab (APDM-sensors) | month 3
  static and dynamic balance using the Mobility lab (APDM-sensors): iSway (COP sway area and velocity with and without vision), iTUG
Four Test Balance Scale (4TBS) | baseline
Four Test Balance Scale (4TBS) | month 1
Four Test Balance Scale (4TBS) | month 2
Four Test Balance Scale (4TBS) | month 3
Four Test Balance Scale (4TBS) | month 4
Four Test Balance Scale (4TBS) | month 5
Four Test Balance Scale (4TBS) | month 6
Functional Ambulation categories (FAC) | baseline
Functional Ambulation categories (FAC) | month 1
Functional Ambulation categories (FAC) | month 2
Functional Ambulation categories (FAC) | month 3
Functional Ambulation categories (FAC) | month 4
Functional Ambulation categories (FAC) | month 5
Functional Ambulation categories (FAC) | month 6
Dizziness Handicap Inventory (DHI) | baseline
Dizziness Handicap Inventory (DHI) | month 3

SECONDARY OUTCOMES:
Fall incidents | baseline
Fall incidents | month 1
Fall incidents | month 2
Fall incidents | month 3
Fall incidents | month 4
Fall incidents | month 5
Fall incidents | month 6
fear of falling | baseline
  fear of falling: Falls Efficacy Scale
fear of falling | month 3
  fear of falling: Falls Efficacy Scale
depression | baseline
  depression: Geriatric depression scale
depression | month 3
  depression: Geriatric depression scale
ambulatory activity level | baseline
  ambulatory activity level: the StepWatch Activity Monitor (SAM)
ambulatory activity level | month 3
  ambulatory activity level: the StepWatch Activity Monitor (SAM)

CONTACTS AND LOCATIONS:
Overall Officials: Joke spildooren, dr., Principal Investigator — Hasselt University
Locations (1):
- Hasselt University, Hasselt, Belgium

IPD SHARING:
Plan to Share IPD: Undecided